CLINICAL TRIAL: NCT06906445
Title: Efficacy of Microbiome Manipulation Strategies Fecal Microbial Transplant or Anti-inflammatory Diet or Both With Advanced Therapies BiOlOgics and Small Molecules to Break the Therapeutic Ceiling in Active Ulcerative Colitis BOOST-UC A Multicenter Double Blind Factorial Randomized Controlled Trial
Brief Title: A Study to Evaluate the Effect of Fecal Transplant and Dietary Changes on Disease Activity in Patients With Ulcerative Colitis on Advanced Therapies
Acronym: BOOST-UC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Prof. Vineet Ahuja, Professor, All India Institute of Medical Sciences
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: AIIMSA2987/03.01.2025; EMDR/CARE/12/2023-0000572 (Other Grant/Funding Number: Indian Council of Medical Research, New Delhi, India)
Record Dates: First submitted 2025-03-03; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Ulcerative Colitis
Keywords: Randomized Controlled Trial; Fecal Microbial Transplantation; Anti-inflammatory diet; Factorial design; Ulcerative colitis; Advanced therapy
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Fecal Microbiota Transplantation and Anti inflammatory diet and advanced therapy (Experimental): 1.Oral vancomycin 500 mg BD for 3 days before the first FMT 2.FMT via colonoscopy at 0, 2, and 6 weeks for induction of remission 3.FMT via colonoscopy every 8 weeks (week 10, 18, 26, 34, 42) for maintenance of remission, if the patient is responder to the induction therapy 4.If the patient is a non-responder or has treatment failure to induction, he/she will be withdrawn from the study. 5.Patients with secondary loss of response, in the maintenance phase, will be withdrawn from the study 6.AID for 48 weeks. 7.Advanced therapy as standard dose and schedule
  Interventions: Other: Fecal Microbial Transplantation; Other: Anti-Inflammatory Diet; Other: Advanced Therapy
- Fecal Microbiota Transplantation and sham diet/standard dietary counselling and advanced therapy (Experimental): 1.Oral vancomycin 500 mg BD for 3 days before the first FMT 2.FMT via colonoscopy at 0, 2, and 6 weeks for induction of remission 3.FMT via colonoscopy every 8 weeks (week 10, 18, 26, 34, 42) for maintenance of remission, if the patient is responder to the induction therapy 4.If the patient is a non-responder or has treatment failure to induction, he/she will be withdrawn from the study. 5.Patients with secondary loss of response, in the maintenance phase, will be withdrawn from the study 6. Sham AID/Standard dietary counseling for 48 weeks. 7. Advanced therapy as standard dose and schedule
  Interventions: Other: Fecal Microbial Transplantation; Other: Sham Diet; Other: Advanced Therapy
- Sham Transplantation and Anti inflammatory diet and advanced therapy (Experimental): 1.Oral placebo 1 BD for 3 days before first FMT 2.Sham FMT via colonoscopy (instillation of clean water) at 0, 2, and 6 weeks 3.Sham FMT via colonoscopy (instillation of clean water) every 8 weeks (week 10, 18, 26, 34, 42) for maintenance of remission, if the patient is responder to the induction therapy 4.If the patient is a non-responder or has treatment failure to induction therapy, he/she will be withdrawn from the study. 5.Patients with secondary loss of response, in the maintenance phase, will be withdrawn from the study 6. AID for 48 weeks. 7. Advanced therapy as standard dose and schedule.
  Interventions: Other: Anti-Inflammatory Diet; Other: Sham transplantation; Other: Advanced Therapy
- Sham transplantation and Sham Diet and advanced therapy (Sham Comparator): 1.Oral placebo 1 BD for 3 days before first FMT 2. Sham FMT via colonoscopy (instillation of clean water) at 0, 2, and 6 weeks 3. Sham FMT via colonoscopy (instillation of clean water) every 8 weeks (week 10, 18, 26, 34, 42) for maintenance of remission, if the patient is responder to the induction therapy 4. If the patient is a non-responder or has treatment failure to induction therapy, he/she will be withdrawn from the study. 5. Patients with secondary loss of response, in the maintenance phase, will be withdrawn from the study 6. Sham AID/Standard dietary counseling for 48 weeks 7. Advanced therapy as standard dose and schedule
  Interventions: Other: Sham transplantation; Other: Sham Diet; Other: Advanced Therapy

INTERVENTIONS:
Other: Fecal Microbial Transplantation — This will involve colonoscopic instillation of fecal transplant
  Arms: Fecal Microbiota Transplantation and Anti inflammatory diet and advanced therapy; Fecal Microbiota Transplantation and sham diet/standard dietary counselling and advanced therapy
Other: Anti-Inflammatory Diet — The modified diet plan will be given to each study participant
  Arms: Fecal Microbiota Transplantation and Anti inflammatory diet and advanced therapy; Sham Transplantation and Anti inflammatory diet and advanced therapy
Other: Sham transplantation — Sham FMT will involve saline infusion via colonoscopy
  Arms: Sham Transplantation and Anti inflammatory diet and advanced therapy; Sham transplantation and Sham Diet and advanced therapy
Other: Sham Diet — Dietary counselling alone
  Arms: Fecal Microbiota Transplantation and sham diet/standard dietary counselling and advanced therapy; Sham transplantation and Sham Diet and advanced therapy
Other: Advanced Therapy — Advanced therapy as standard dose and schedule

SUMMARY:
Ulcerative colitis (UC) is a chronic inflammatory disease of the colon characterized by superficial mucosal inflammation. Treatment aims to achieve and maintain remission, improve quality of life, and minimize complications. Advanced therapies, including biologics and small molecules, have significantly improved UC management by targeting specific inflammatory pathways. However, due to the multifactorial nature of UC-driven by genetic, environmental, and microbial factors-many patients do not achieve sustained remission, highlighting a therapeutic ceiling. Gut microbial dysbiosis and immune dysregulation are central to UC pathogenesis, with diet playing a critical role in influencing the gut microbiome. While biologics and small molecules have limitations, innovative approaches like combining fecal microbiota transplantation (FMT) and dietary interventions with advanced therapies show promise. FMT restores microbial balance, modulates immunity, and reduces inflammation, while dietary modifications, such as anti-inflammatory diets, enhance FMT efficacy by creating a favorable environment for donor microbiota engraftment. The present study is designed to evaluate the efficacy of three different microbiome manipulation strategies- FMT, AID and FMT + AID in combination with advanced therapies in patients with active UC in a 2X2 factorial trial design. Patients would be randomized into four different arms: FMT, AID, FMT+AID and placebo. The advanced therapies (biologics or small molecules) would be given in all four arms as standard therapy. With this design the trial would answer two important questions: a) efficacy of combination treatment with advanced therapies and microbiome manipulation strategies in active UC, and b) comparative efficacy of different microbiome manipulation strategies.

DETAILED DESCRIPTION:
This study is a multicenter, randomized, factorial-design, double-blind, controlled trial investigating the effects of fecal microbiota transplantation (FMT) and dietary interventions in patients with mild to moderate, treatment-naïve, active inflammatory bowel disease. The trial is being conducted across multiple clinical centers, with a central microbiome analysis facility.

Randomization and Blinding:

Randomization: Centralized, computerized randomization is employed to ensure balanced treatment allocation. The permuted block method, along with stratification based on disease characteristics, ensures equal distribution across intervention arms Blinding: Patients, investigators collecting clinical data, and endoscopic video assessors are blinded to treatment allocation. The dietitian and endoscopist performing FMT (or sham FMT) are unblinded

Intervention Arms:

Participants are assigned to one of four treatment arms:

FMT + Anti-inflammatory Diet (AID) +Advanced therapy FMT + Sham Diet+ Advanced therapy Sham FMT + AID+ Advanced therapy Sham FMT + Sham Diet+ Advanced therapy FMT is administered via colonoscopy at 0, 2, and 6 weeks, with responders receiving maintenance doses every 8 weeks until week 48

Participant Timeline and Assessments:

Baseline Assessments: Clinical, laboratory, and endoscopic evaluations, including serological tests, inflammatory markers, and microbiome profiling.

Follow-up Schedule: Visits occur at Week 0, Week 6, Week 10, and then every 8 weeks until Week 48.

Endoscopic Monitoring: Colonoscopy is performed at baseline, Week 10, and Week 48. Centralized endoscopic video scoring ensures consistency

Data Collection and Management:

Paper CRF's and Electronic Data: The paper based CRF's will be filled first and then data will be entered into a REDCap software.

Dietary Monitoring: Participants will use the IBD NutriCare mobile application for diet tracking.

Microbiome Analysis: Fecal samples are processed and analyzed at a designated microbiome research center.

Safety Monitoring and Compliance:

Adverse Event Reporting: All safety events, including potential serious adverse events (SAEs), are logged and monitored by the Data and Safety Monitoring Board (DSMB).

Protocol Deviations: Documented and assessed for impact on trial integrity. Training and Quality Control: Regular site training ensures adherence to the protocol, and periodic audits maintain data quality

ELIGIBILITY:
Inclusion Criteria:

1. Adult (age 18 to 75 years) patients
2. Patients with active UC (defined as mMS equal or greater than 3 with rectal bleed score equal or greater than 1 and Endoscopic Mayo score equal or greater than 2 documented within 3 months of randomization or mild symptoms with high inflammatory burden or poor prognostic features).
3. Any disease extent E1, E2 or E3. Patients with Proctitis will be limited to 25 percent of the entire pool of patients.
4. Patients with an inadequate response, loss of response, or intolerance to conventional therapies example, aminosalicylates, corticosteroids, immunosuppressants or advanced therapies including but not limited to anti TNF alpha agents, anti-integrins, anti IL 12 or IL 23 agents, anti IL 23 agents, JAK inhibitors, or S1P receptor modulators. The last administration of any such treatment must have occurred at least five half-lives prior to randomization.
5. Confirmed diagnosis of UC. The diagnosis must be confirmed by endoscopic and histologic evidence and corroborated by a histopathology report
6. Subjects who are willing and able to comply with treatment plan, laboratory tests, daily bowel movement diary call and other study procedures
7. Subjects who are willing to provide a written informed consent for FMT
8. Agree to adhere to the diet schedule
9. Infective colitis ruled out Biopsy showing crypt architecture distortion or basal plasmacytosis, OR two sigmoidoscopies, at least 7 days apart showing evidence of endoscopic activity

Exclusion Criteria:

1. Hospitalization of exacerbation of UC requiring intravenous corticosteroids
2. Patients already on biologics (anti-tumor necrosis factor inhibitors) or small molecules (tofacitinib) for equal or more than 2 weeks.
3. Clinical signs of fulminant colitis or toxic megacolon
4. Positive assay or stool culture for pathogens (ova and parasite examination, bacteria) or positive test for Clostridioides difficile toxin or CMV (histology or IHC and or tissue PCR) at screening. (The patients with positive assay will be treated appropriately and tests will be repeated. Those with negative assay and persistent activity will be included in the study.)
5. Active or inadequately treated infections, including Mycobacterium tuberculosis.
6. Presence of IBD-unclassified, microscopic colitis, ischemic colitis, infectious colitis, or clinical findings suggestive of Crohn's Disease.
7. Patients infected with human immunodeficiency virus (HIV)
8. Patients with current or past history of malignancy.
9. Patients with current or recent history of clinically severe, progressive, or uncontrolled renal, hepatic, Hematological, gastrointestinal, metabolic, endocrine, pulmonary, cardiac, or neurological disease.
10. Pregnant females

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-03-15 (Actual); Primary Completion 2027-03-15 (Estimated); Study Completion 2028-03-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of Patients Achieving Clinical Remission and Endoscopic Response at 10 weeks | 10 weeks
  Proportion of patients having- 1. Clinical remission which is defined as the Modified Mayo Score (mMS) < 2 \ mMS- Full Title: Modified Mayo Score Range: 0 to 12 Higher Scores = Worse Outcome (A score of 0 represents no disease activity, and a score of 12 represents the most severe disease activity.) 2. Endoscopic response which is defined as Mayo Endoscopic Score (MES) by 1 point MES- Full Title: Mayo Endoscopic Score Range: 0 to 4 Higher Scores = Worse Outcome (A score of 0 represents normal endoscopic findings, and a score of 4 represents severe mucosal damage.
Proportion of patients having clinical remission and endoscopic remission at week 48 | 48 weeks
  Proportion of patients having- 1. Clinical remission which is defined as the Modified Mayo Score (mMS) < 2 mMS- Full Title: Modified Mayo Score Range: 0 to 12 Higher Scores = Worse Outcome (A score of 0 represents no disease activity, and a score of 12 represents the most severe disease activity.) 2. Endoscopic response which is defined as Mayo Endoscopic Score (MES) by 1 point MES- Full Title: Mayo Endoscopic Score Range: 0 to 4 Higher Scores = Worse Outcome (A score of 0 represents normal endoscopic findings, and a score of 4 represents severe mucosal damage.

SECONDARY OUTCOMES:
Proportion of patients having clinical response at week 10 | 10 weeks
  Proportion of patients having clinical response (Defined as a decrease from baseline in the mMS of greater than or equal to 2 points and at least a 30 percent reduction from baseline) mMS- Full Title: Modified Mayo Score Range: 0 to 12 Higher Scores = Worse Outcome (A score of 0 represents no disease activity, and a score of 12 represents the most severe disease activity.)
Proportion of patients having clinical remission at week 10 | 10 weeks
  Proportion of patients having clinical remission which is defined as an mMS of 0 to 2, including the following three components: 1) Stool frequency sub score = 0 (or = 1 with a ≥ 1-point decrease from baseline), 2) Rectal bleeding sub score = 0 3) Centrally read endoscopy sub score = 0 or 1 (score of 1 modified to exclude friability) mMS- Full Title: Modified Mayo Score Range: 0 to 12 Higher Scores = Worse Outcome (A score of 0 represents no disease activity, and a score of 12 represents the most severe disease activity.)
Proportion of Patients achieving Symptomatic Response at Week 10 | 10 weeks
  Proportion of Patients Achieving Symptomatic Response which is defined as Decrease from baseline ≥ 30% in composite Rectal Bleeding sub score and Stool Frequency sub score and a ≥ 1-point decrease from baseline in RB sub score or an absolute RB sub score ≤ 1) Stool Frequency Subscore: Range: 0 to 3 (typically; the exact range may vary depending on the scale used) Lower Scores = Better Outcome (A score of 0 indicates no stool frequency issues, while higher scores represent increasing frequency of stools, indicating worse disease activity.) Rectal Bleeding Subscore: Range: 0 to 3 (typically; range may vary depending on the version used) Lower Scores = Better Outcome (A score of 0 indicates no rectal bleeding, while higher scores represent increasing severity of rectal bleeding, indicating worse disease activity.)
Proportion of Patients achieving Symptomatic Remission at week 10 | 10 weeks
  Proportion of Patients achieving Symptomatic Remission which is defined as Stool Frequency subscore = 0 (or = 1 with a ≥ 1-point decrease from baseline) and Rectal Bleeding subscore = 0 Stool Frequency Subscore: Range: 0 to 3, Lower Scores = Better Outcome (A score of 0 indicates no stool frequency issues, while higher scores represent increasing frequency of stools, indicating worse disease activity.) Rectal Bleeding Subscore: Range: 0 to 3, Lower Scores = Better Outcome (A score of 0 indicates no rectal bleeding, while higher scores represent increasing severity of rectal bleeding, indicating worse disease disease activity.) Rectal Bleeding Subscore: Range: 0 to 3, Lower Scores = Better Outcome (A score of 0 indicates no rectal bleeding, while higher scores represent increasing severity of rectal bleeding, indicating worse disease activity.)
Proportion of Patients Achieving Endoscopic Response at Week 10 | 10 weeks
  Proportion of Patients Achieving Endoscopic Response which is defined as decrease in Modified Endoscopic Score ≥1 points MES- Full Title: Mayo Endoscopic Score Range: 0 to 4 Higher Scores = Worse Outcome (A score of 0 represents normal endoscopic findings, and a score of 4 represents severe mucosal damage.
Proportion of Patients Achieving Endoscopic Remission at Week 10 | 10 weeks
  Proportion of Patients achieving Endoscopic Remission which is defined as Modified Endoscopy Score=0 MES- Full Title: Mayo Endoscopic Score Range: 0 to 4 Higher Scores = Worse Outcome (A score of 0 represents normal endoscopic findings, and a score of 4 represents severe mucosal damage.
Proportion of Patients Achieving Histologic Remission at Week 10 | 10 weeks
  Proportion of Patients Achieving Histologic Remission (Robarts histopathology index score <3 with lamina propria neutrophils score = 0 and neutrophil in epithelium score=0; DCA (Distribution/ chronicity/ activity) score, A=0) Robarts Histopathology Index (RHI): Full Title: Robarts Histopathology Index Range: 0 to 16 (varies depending on the specific version used, but typically it is in this range) Lower Scores = Better Outcome (A lower score indicates less histologic damage or inflammation.) Lamina Propria Neutrophils Score: Range: 0 to 3 Lower Scores = Better Outcome (A score of 0 indicates no neutrophils present, which is a sign of histologic remission.) Neutrophils in Epithelium Score: Range: 0 to 3 Lower Scores = Better Outcome (A score of 0 indicates no neutrophils in the epithelium, which is also a sign of histologic remission.) DCA Score: Full Title: Distribution/Chronicity/Activity Score Range: 0 to 3 Lower Scores = Better Outcome (score of 0 =no activity
Proportion of Patients Achieving Biomarker Remission at Week 10 | 10 weeks
  Proportion of Patients Achieving Biomarker Remission (Defined as fecal calprotectin ≤150 mcg/g) at Week 10
Proportion of Patients Experiencing Adverse Events at Week 10 | 10 weeks
  Proportion of Patients experiencing Adverse events which will be assessed according to the Common Terminology Criteria for Adverse Events (CTCAE) and graded as follows: Grade 1: Mild symptoms (no intervention required). Grade 2: Moderate symptoms (non-operative intervention required). Grade 3: Severe symptoms (operative intervention required). Grade 4: Life-threatening consequences (urgent intervention required). Grade 5: Death.
Fecal Microbiome and Metabolite Signature at Week 10 | 10 weeks
  It involves combined analysis of the microorganisms (bacteria, viruses, fungi, etc.) and the small molecules (metabolites) present in a person's stool sample
Dynamics of microbiome engraftment at week 10 | 10 weeks
  It involves capturing donor-to-recipient microbiome transfer/shift at species and strain-level will be performed as an investigation of 'FMT events', where in each event will include triad of samples: the donor, the Pre-FMT and the Post-FMT sample from the recipient patient. Species-level donor-to-recipient shifts will be investigated by computing the Bray-Curtis and Kendall distances between all three sample-pairs of the triad. Kendall distances capture the variations and similarities amongst samples in terms of the relative hierarchical ranking of different taxa within a community, Bray-Curtis distances capture the differences in the abundances of different taxa across two communities. Both these distance measure-based approaches will be utilized the fraction of recipient microbiome that is modulated by the donor microbiome in terms of both composition and species-level hierarchy.
Proportion of patients having clinical response at week 48 | 48 weeks
  Proportion of patients having clinical response (Defined as a decrease from baseline in the mMS of greater than or equal to 2 points and at least a 30 percent reduction from baseline) mMS- Full Title: Modified Mayo Score Range: 0 to 12 Higher Scores = Worse Outcome (A score of 0 represents no disease activity, and a score of 12 represents the most severe disease activity.)
Proportion of patients having clinical remission at week 48 | 48 weeks
  Proportion of patients having clinical remission which is defined as an modified mayo score of 0 to 2, including the following three components: 1) Stool frequency sub score = 0 (or = 1 with a ≥ 1-point decrease from baseline), 2) Rectal bleeding sub score = 0 3) Centrally read endoscopy sub score = 0 or 1 (score of 1 modified to exclude friability) mMS- Full Title: Modified Mayo Score Range: 0 to 12 Higher Scores = Worse Outcome (A score of 0 represents no disease activity, and a score of 12 represents the most severe disease activity.)
Proportion of Patients Achieving Symptomatic Response at Week 48 | 48 weeks
  Proportion of Patients Achieving Symptomatic Response which is defined as Decrease from baseline ≥ 30% in composite Rectal Bleeding sub score and Stool Frequency sub score and a ≥ 1-point decrease from baseline in RB sub score or an absolute RB sub score ≤ 1) Stool Frequency Subscore: Range: 0 to 3 (typically; the exact range may vary depending on the scale used) Lower Scores = Better Outcome (A score of 0 indicates no stool frequency issues, while higher scores represent increasing frequency of stools, indicating worse disease activity.) Rectal Bleeding Subscore: Range: 0 to 3 (typically; range may vary depending on the version used) Lower Scores = Better Outcome (A score of 0 indicates no rectal bleeding, while higher scores represent increasing severity of rectal bleeding, indicating worse disease activity.)
Proportion of Patients achieving Symptomatic Remission at Week 48 | 48 weeks
  Proportion of Patients achieving Symptomatic Remission which is defined as Stool Frequency subscore = 0 (or = 1 with a ≥ 1-point decrease from baseline) and Rectal Bleeding subscore = 0 Stool Frequency Subscore: Range: 0 to 3 (typically; the exact range may vary depending on the scale used) Lower Scores = Better Outcome (A score of 0 indicates no stool frequency issues, while higher scores represent increasing frequency of stools, indicating worse disease activity.) Rectal Bleeding Subscore: Range: 0 to 3 (typically; range may vary depending on the version used) Lower Scores = Better Outcome (A score of 0 indicates no rectal bleeding, while higher scores represent increasing severity of rectal bleeding, indicating worse disease activity.)
Proportion of Patients achieving Endoscopic Response at Week 48 | 48 weeks
  Proportion of Patients Achieving Endoscopic Response which is defined as decrease in Modified Endoscopic Score ≥1 points MES- Full Title: Mayo Endoscopic Score Range: 0 to 4 Higher Scores = Worse Outcome (A score of 0 represents normal endoscopic findings, and a score of 4 represents severe mucosal damage.
Proportion of Patients achieving Endoscopic Remission at Week 48 | 48 weeks
  Proportion of Patients achieving Endoscopic Remission which is defined as Modified Endoscopy Score=0 MES- Full Title: Mayo Endoscopic Score Range: 0 to 4 Higher Scores = Worse Outcome (A score of 0 represents normal endoscopic findings, and a score of 4 represents severe mucosal damage.
Proportion of Patients achieving Histologic Remission at Week 48 | 48 weeks
  Proportion of Patients Achieving Histologic Remission (Robarts histopathology index score <3 with lamina propria neutrophils score = 0 and neutrophil in epithelium score=0; DCA (Distribution/ chronicity/ activity) score, A=0) Robarts Histopathology Index (RHI): Full Title: Robarts Histopathology Index Range: 0 to 16 (varies depending on the specific version used, but typically it is in this range) Lower Scores = Better Outcome (A lower score indicates less histologic damage or inflammation.) Lamina Propria Neutrophils Score: Range: 0 to 3 Lower Scores = Better Outcome (A score of 0 indicates no neutrophils present, which is a sign of histologic remission.) Neutrophils in Epithelium Score: Range: 0 to 3 Lower Scores = Better Outcome (A score of 0 indicates no neutrophils in the epithelium, which is also a sign of histologic remission.) DCA Score: Full Title: Distribution/Chronicity/Activity Score Range: 0 to 3 Lower Scores = Better Outcome (score of 0 =no activity
Proportion of Patients Achieving Biomarker Remission at Week 48 | 48 weeks
  Proportion of Patients Achieving Biomarker Remission (Defined as fecal calprotectin ≤150 mcg/g)
Fecal Microbiome and Metabolite Signature at Week 48 | 48 weeks
  It involves combined analysis of the microorganisms (bacteria, viruses, fungi, etc.) and the small molecules (metabolites) present in a person's stool sample
Dynamics of microbiome engraftment at week 48 | 48 weeks
  It involves capturing donor-to-recipient microbiome transfer/shift at species and strain-level will be performed as an investigation of 'FMT events', where in each event will include triad of samples: the donor, the Pre-FMT and the Post-FMT sample from the recipient patient. Species-level donor-to-recipient shifts will be investigated by computing the Bray-Curtis and Kendall distances between all three sample-pairs of the triad. Kendall distances capture the variations and similarities amongst samples in terms of the relative hierarchical ranking of different taxa within a community, Bray-Curtis distances capture the differences in the abundances of different taxa across two communities. Both these distance measure-based approaches will be utilized the fraction of recipient microbiome that is modulated by the donor microbiome in terms of both composition and species-level hierarchy.
Proportion of Patients Experiencing Adverse Events at Week 48 | 48 weeks
  Proportion of Patients experiencing Adverse events which will be assessed according to the Common Terminology Criteria for Adverse Events (CTCAE) and graded as follows: Grade 1: Mild symptoms (no intervention required). Grade 2: Moderate symptoms (non-operative intervention required). Grade 3: Severe symptoms (operative intervention required). Grade 4: Life-threatening consequences (urgent intervention required). Grade 5: Death.
Proportion of patients having adverse events at week 6 | 6 weeks
  Proportion of Patients experiencing Adverse events which will be assessed according to the Common Terminology Criteria for Adverse Events (CTCAE) and graded as follows: Grade 1: Mild symptoms (no intervention required). Grade 2: Moderate symptoms (non-operative intervention required). Grade 3: Severe symptoms (operative intervention required). Grade 4: Life-threatening consequences (urgent intervention required). Grade 5: Death.
Proportion of patients having adverse events at week 26 | 26 weeks
  Proportion of Patients experiencing Adverse events which will be assessed according to the Common Terminology Criteria for Adverse Events (CTCAE) and graded as follows: Grade 1: Mild symptoms (no intervention required). Grade 2: Moderate symptoms (non-operative intervention required). Grade 3: Severe symptoms (operative intervention required). Grade 4: Life-threatening consequences (urgent intervention required). Grade 5: Death.

CONTACTS AND LOCATIONS:
Overall Officials: Prof Vineet Ahuja, DM Gastroenterology, Principal Investigator — Department of Gastroenterology, AIIMS, New Delhi
Locations (6):
- India (6):
  - Department of Gastroenterology, Lisie Hospital, Kochi, Kerala
  - Lokmanya Tilak Municipal General Hospital and Lokmanya Tilak Municipal Medical College, Sion, Mumbai, Maharashtra
  - Department of Gastroenterology and Human Nutrition, All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi
  - Department of Gastroenterology, Dayanand Medical College, Ludhiana, Punjab
  - Department of Gastroentrology, Postgraduate Institute of Medical Education and Research,, Chandigarh, Punjab/Haryana
  - Department of Gastroenterology, Institute of Medical Sciences, Varanasi, Uttar Pradesh

IPD SHARING:
Plan to Share IPD: No